CLINICAL TRIAL: NCT03549676
Title: Fecal Microbiota Transplantation for Treatment of Refractory Graft Versus Host Disease-a Pilot Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Cao Qing, Director of Infectious Diseases, Shanghai Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-GVHD
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Fecal Microbiota Transplantation in GVHD
Keywords: FMT; GVHD; HSCT
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSCT patients with refractory GVHD (Experimental): Patients will accept FilmArray Gastrointestinal (GI) panel test before pre-treatment of HSCT and 28±3 days post-HSCT. Patients will receive 50ml fecal microbiota from unrelated healthy donors through nasojejunal tube and monitored under gastroscopy. Patients receiving FMT treatment will be followed for at least 6 months. The ideal follow up time is 2 year. Stool and blood samples will be serially collected and tested (before pre-treatment, 1/3/6/12 months after FMT).
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — For patients who do not respond or partial respond for first time FMT treatment, a second time FMT treatment using different donor should be considered.

SUMMARY:
The study evaluates safety and efficacy of fecal microbiota transplantation (FMT) for the treatment of refractory graft-versus-host-disease (GVHD) of the gut. FMT might be a beneficial treatment in this clinical situation with a poor prognosis and limited therapeutic options.

DETAILED DESCRIPTION:
Graft-versus-host-disease (GVHD) is a major complication after hematopoietic stem cell transplantation (HSCT). Gut is the most vulnerable target organ of acute GVHD. Patients who have a gastrointestinal acute GVHD received a first-line standard treatment of corticosteroids. For patients who do not respond or progress after an initial response have a high mortality. Therefore, the investigation of effective second line therapy for these patients are in need. The study evaluates safety and efficacy of fecal microbiota transplantation (FMT) for the treatment of refractory GVHD of the gut. FMT might be a beneficial treatment in this clinical situation with a poor prognosis and limited therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* 3-18 years of age
* Allo-SCT patients with acute steroid-resistant GI-related GVHD grade III-IV. Steroid-resistant GI-related GVHD will be defined as lack of improvement (same stage) or worsening of GI symptoms after 7 days of steroid therapy (≥ 2 ml/kg of IV methylprednisolone)
* No definite contraindication for gastrointestinal endoscopy
* Signature of informed consent by the legal guardians of patients

Exclusion Criteria:

* Prior inclusion to an interventional study
* Previous Allo-SCT
* Known multi-drug resistance carriage prior to stool collection
* Severe colitis of any etiology or a history of inflammatory bowel disease (IBD)
* Uncontrolled infection (hemodynamic instability, ongoing high fever or bacteremia within 3 days after antibiotics administration)
* Active GI bleeding
* Absolute neutrophil count < 500 cells/microL
* Absolute platelet count< 10 x 109 /L
* Patients who cannot give informed consent

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of FMT in the treatment of refractory GVHD on day 7 | 7 days following FMT
  Participants will be evaluated on days 7 following FMT. The volume and frequency of daily diarrhoea will be continuous observed and recorded in 7 days.
Efficacy of FMT in the treatment of refractory GVHD on day 28 | 28 days following FMT
  Participants will be evaluated on days 28 following FMT. The volume and frequency of daily diarrhoea will be continuous observed and recorded in 28 days.

SECONDARY OUTCOMES:
Treatment-related AEs and SAEs | up to 28 days following FMT
  The overall safety of the study will be evaluated with the incidence of all Adverse Events (AEs) and Serious Adverse Events (SAEs) within 28 days following FMT. The relationship of any kind AEs and FMT will be seriously evaluated. Non-serious AEs include: dyspepsia, abdominal pain, nausea, vomiting, diarrhea, constipation, fever, inhalation without mechanical ventilation, etc. SAEs include: death, sepsis, aspiration pneumonia, gastrointestinal hemorrhage, septic shock, etc.
GVHD severity | up to 28 days following FMT
  Patients will be evaluated on days 7 and 28 following transplantation for severity of GVHD. GVHD severity is graded by the International Bone Marrow Transplant Registry Severity Index grading system.
Implantation rate | through study completion, an average of 6 months
  The data will be compared with patients who had not participated in clinical trials.
Survival rate | through study completion, an average of 6 months
  The data will be compared with patients who had not participated in clinical trials.
Change in biomarkers | up to 28 days following FMT
  Change in levels of albumin and C-reactive protein between days 0 and days 28 will serve as a secondary endpoint.
Number of patients with infectious disorders | through study completion, an average of 6 months
  Evaluation of FMT activity on infectious disorder.
Quality of Life | up to 6 months following FMT
  The quality of life of patients will be measured using a standardized quality of life questionnaire (EORTC QLQ-C30) prior to transplantation and on days 7, 14, 21, 28 and 180 following transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Cao, MD, Study Director — Shanghai Children's Medical Center

IPD SHARING:
Plan to Share IPD: Undecided